CLINICAL TRIAL: NCT06786377
Title: Genetic and Clinical Characterization of Type 1 and 2 Narcolepsy in Adult and Pediatric Black and North African Populations
Acronym: NarcoGen
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240964; IDRCB: 2024-A02078-39 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- narcolepsy patients: 50 narcolepsy patients will be included in the study at Robert Debré Hospital
  Interventions: Genetic: saliva sampling
- control patients: 150 control patients will be included in the study at Robert Debré Hospital
  Interventions: Genetic: saliva sampling

INTERVENTIONS:
Genetic: saliva sampling — saliva sampling

SUMMARY:
Narcolepsy type 1 (NT1) is a neurological disorder characterized by excessive daytime sleepiness, cataplexy, sleep paralysis, and hallucinations while awake. It results from the loss of orexin-producing neurons in the hypothalamus, leading to a deficiency of the neuropeptide orexin/hypocretin. Studies show differences in the clinical presentation of NT1 between Caucasian and African American populations, highlighting the importance of research into genetic and clinical characteristics specific to Black and North African populations.

A genetic study in these populations could identify novel genes associated with NT1 and NT2, providing crucial information for personalized diagnosis and treatment. This would fill a knowledge gap and promote more effective interventions for individuals of African descent, contributing to a better understanding of narcolepsy globally.

DETAILED DESCRIPTION:
Narcolepsy type 1 (NT1) is a neurological disease characterized by excessive daytime sleepiness (EDS), cataplexy, sleep paralysis and hypnagogic hallucinations. It is caused by the loss of neurons located in the lateral hypothalamus leading to a sudden deficiency of a neuropeptide hypocretin/orexin involved in the functions of sleep and wakefulness but also food intake and metabolism. NT1 is diagnosed by the presence of EDS and cataplexies or in the absence of cataplexies but with documented hypocretin/orexin deficiency measured in the cerebrospinal fluid (CSF). Other cases without cataplexy (and without orexin deficiency) are classified as narcolepsy type 2 (NT2).

Although narcolepsy has been widely studied in different populations, there is a lack of knowledge about the genetic and clinical characteristics of people of Black and North African descent.

In Caucasian populations, NT1 is associated with specific major histocompatibility complex (MHC) alleles, particularly HLA-DQB1*06:029. However, recent observations in African American populations have indicated a different clinical presentation. Notably, earlier onset, increased prevalence of atypical symptoms, greater prevalence of narcolepsy without cataplexy, and low cerebrospinal fluid orexin levels have been reported. Specifically, the DQB103:01 allele has been associated with NT1 in African Americans. Additionally, in African populations, a specific mutation called DQB103:19 has been identified within the DQB103:0112 allele.

Genome-wide association studies (GWAS) have proven to be of major interest in identifying genetic variations associated with complex disorders. However, the majority of GWAS on narcolepsy have focused on non-African populations. Carrying out a GWAS in black and North African populations is able to provide new information on the genetic architecture of NT1 and NT2 and highlight specific risk factors in this particularly exposed population.

In conclusion, better understanding the genetic and clinical heterogeneity of NT1 and NT2 in black and North African populations is crucial to advance our knowledge of this disease and adapt targeted diagnostic and therapeutic approaches to specific populations. The present study aims to contribute significantly to the understanding of pediatric and adult narcolepsy and to facilitate more personalized and effective interventions for individuals of African descent.

Although narcolepsy has been widely studied in different populations, there is a lack of knowledge about the genetic and clinical characteristics of people of Black and North African descent.

ELIGIBILITY:
Inclusion Criteria:

Narcolepsy patients:

* Individuals of black and North African origin diagnosed with NT1 or NT2.
* Age ≥ 6 years
* Clinical confirmation of narcolepsy according to the criteria of the International Classification of Sleep Disorders (ICSD-3).
* Signature of informed consent by the adult patient or both holders of parental authority for minor patients.

Control subjects:

* Volunteers without pathology related to the study from the same ethnic or related groups with the aim of reaching two matched control subjects for each case.
* Age ≥ 6 years
* Signature of informed consent by the adult subject or both holders of parental authority for minor subjects.

Exclusion Criteria:

* Individuals unable to understand the protocol or unwilling to participate.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Narcolepsy patients with NT1 or NT2.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Describe the genetic and clinical features of type 1 and 2 narcolepsy in Black and North African populations | 12 months
  Presence of genetic specificity in the populations studied

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided